CLINICAL TRIAL: NCT01653470
Title: A Phase Ib Ascending Multi-arm, Dose Escalation Study of BMS-906024 Combined With Several Chemotherapy Regimens in Subjects With Advanced or Metastatic Tumors
Brief Title: Study to Evaluate Safety & Tolerability of BMS-906024 in Combination With Chemotherapy & to Define DLTs & MTD of BMS-906024 in Combination With One of the Following Chemotherapy Regimens; Weekly Paclitaxel, 5FU+Irinotecan or Carboplatin+Paclitaxel in Subjects With Advanced / Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA216-003; 2012-003232-23 (EudraCT Number)
Record Dates: First submitted 2012-07-18; First posted 2012-07-31 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Paclitaxel; Fluorouracil; Carboplatin; Leucovorin; Irinotecan; BMS-906024

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A: Paclitaxel + BMS-906024 (Experimental): Paclitaxel 80 mg/m2 solution and BMS-906024 4 mg or 6 mg solution intravenously once weekly continuously until disease progression or unacceptable toxicity
  Interventions: Drug: Paclitaxel; Drug: BMS-906024
- Arm B: FOLFIRI (5FU, Leucovorin, Irinotecan) + BMS-906024 (Experimental): 5FU Bolus 400 mg/m2, 5FU Infusion 2400 mg/m2, Irinotecan 180 mg/m2 solution, Leucovorin 400 mg/m2 solution intravenously once every 2 weeks and BMS- 906024 4 mg or 6 mg solution intravenously once weekly continuously until disease progression or unacceptable toxicity
  Interventions: Drug: 5-Fluorouracil (5FU); Drug: Leucovorin; Drug: Irinotecan; Drug: BMS-906024
- Arm C: Carboplatin/Paclitaxel + BMS-906024 (Experimental): Carboplatin AUC 6 / Paclitaxel 200 mg/m2 solution once every 3 weeks and BMS-906024 4 mg or 6 mg solution once weekly intravenously continuously until disease progression or unacceptable toxicity
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: BMS-906024
- Arm D: Paclitaxel + BMS-906024 (Experimental): Paclitaxel 80 mg/m2 solution once weekly and BMS-906024 4 mg or 6 mg solution once every 2 weeks intravenously continuously until disease progression or unacceptable toxicity
  Interventions: Drug: Paclitaxel; Drug: BMS-906024
- Arm F: Carboplatin/Paclitaxcel and BMS-906024 (Experimental): Carboplatin AUC 6 / Paclitaxel 200 mg/m2 solution once every 3 weeks and BMS-906024 4 mg or 6 mg solution once every 3 weeks intravenously continuously until disease progression or unacceptable toxicity
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: BMS-906024

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: Taxol
  Arms: Arm A: Paclitaxel + BMS-906024
Drug: 5-Fluorouracil (5FU)
  Other Names: Adrucil; Carac; Efudix; Efudex; Fluoroplex
  Arms: Arm B: FOLFIRI (5FU, Leucovorin, Irinotecan) + BMS-906024
Drug: Carboplatin
  Other Names: Paraplatin
  Arms: Arm C: Carboplatin/Paclitaxel + BMS-906024; Arm F: Carboplatin/Paclitaxcel and BMS-906024
Drug: Leucovorin
  Arms: Arm B: FOLFIRI (5FU, Leucovorin, Irinotecan) + BMS-906024
Drug: Irinotecan
  Other Names: Camptosar
  Arms: Arm B: FOLFIRI (5FU, Leucovorin, Irinotecan) + BMS-906024
Drug: Paclitaxel
  Other Names: Taxol
  Arms: Arm C: Carboplatin/Paclitaxel + BMS-906024; Arm D: Paclitaxel + BMS-906024; Arm F: Carboplatin/Paclitaxcel and BMS-906024
Drug: BMS-906024
  Other Names: Notch inhibitor

SUMMARY:
The purpose of this study is to identify a safe and tolerable dose of BMS-906024 in combination with each of the following three chemotherapy regimens: Paclitaxel, 5FU plus Irinotecan (FOLFIRI), or Carboplatin plus Paclitaxel in subjects with advanced or metastatic solid tumors

DETAILED DESCRIPTION:
DLTs = dose-limiting toxicities

MTD = Maximum tolerated dose

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Subjects with advanced or metastatic solid tumors for whom a chemotherapy regimen is considered appropriate
* Subjects with non-small cell lung cancer and triple-negative breast cancer are preferred
* Biopsy accessible tumor (may use archived tumor samples under certain circumstances)
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Measurable disease

Exclusion Criteria:

* Uncontrolled brain metastases
* Infection
* Gastrointestinal (GI) disease with increased risk of diarrhea (e.g. inflammatory bowel disease)
* Uncontrolled or significant cardiovascular disease
* Subjects taking medications known to increase risk of Torsades de Pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-10-12 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Safety assessment based on reports of adverse events and clinical laboratory tests as graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) | Up to 30 days after the last dose of study medication

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-906024 and BMS-911557 (the active metabolite of BMS-906024), Paclitaxel, Irinotecan, SN-38 (the active metabolite of Irinotecan) and Carboplatin | 16 time points up to first 3 cycles
  Duration of first 3 cycles for Arm A: 10 weeks; Arm B: 6 weeks; Arm C: 9 weeks
Trough observed plasma concentration (Cmin) of BMS-906024 and BMS-911557 (the active metabolite of BMS-906024), Paclitaxel, Irinotecan, SN-38 (the active metabolite of Irinotecan) and Carboplatin | 16 time points up to first 3 cycles
  Duration of first 3 cycles for Arm A: 10 weeks; Arm B: 6 weeks; Arm C: 9 weeks
Time of maximum observed plasma concentration (Tmax) of BMS-906024 and BMS-911557 (the active metabolite of BMS-906024), Paclitaxel, Irinotecan, SN-38 (the active metabolite of Irinotecan) and Carboplatin | 16 time points up to first 3 cycles
  Duration of first 3 cycles for Arm A: 10 weeks; Arm B: 6 weeks; Arm C: 9 weeks
Area under the concentration-time curve during a dosing interval of tau [AUC(TAU)] of BMS-906024 and BMS-911557 (the active metabolite of BMS-906024) | 16 time points up to first 3 cycles
  Duration of first 3 cycles for Arm A: 10 weeks; Arm B: 6 weeks; Arm C: 9 weeks
Area under the concentration-time curve from time 0 to the time of the last sample collected in the dosing interval [AUC(0-T)] of Paclitaxel, Irinotecan, SN-38 (the active metabolite of Irinotecan) and Carboplatin | 16 time points up to first 3 cycles
  Duration of first 3 cycles for Arm A: 10 weeks; Arm B: 6 weeks; Arm C: 9 weeks
Steady-state infusion concentration (Css) of 5-Fluorouracil (5-FU) | 16 time points up to first 3 cycles
  Duration of first 3 cycles for Arm A: 10 weeks; Arm B: 6 weeks; Arm C: 9 weeks
Tumor response [as defined by Response Evaluation Criteria in Solid Tumors (RECIST) (v.1.1) criteria], best overall response (BOR), duration of response, and progression free survival (PFS) will be assessed | Every 6 weeks until confirmed disease progression, death or discontinuation for other reasons (whichever comes first) [Approximately 24 months]
Gene mutation status of Notch activation markers as well as other genes of interest in relevant indications, in tumor, and gene expression levels of Notch activation markers, such as but not limited to Hes1, Deltex1, in tumor | Baseline (study days -28 to -1)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- Usc/Norris Comprehensive Cancer Center, Los Angeles, California, United States
- Local Institution, Brussels, Belgium
- Canada (3):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Toronto, Ontario
  - Local Institution, Ottawa, Quebec

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm